CLINICAL TRIAL: NCT05930483
Title: Using a SMART Design to Evaluate Remotely Delivered, Community-aligned Weight Loss Interventions Among Breast Cancer Survivors: The ¡Vida! Study
Brief Title: Remotely Delivered, Community-Aligned Weight Loss Interventions Among Breast Cancer Survivors, ¡Vida! Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RG1123416; NCI-2023-03748 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0020054 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA270441 (NIH)
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A - Stage 1: ¡Vida!; Stage 2: ¡Vida! (Experimental): Participants participate in the online ¡Vida! program consisting of 24 health education online sessions, dietary modifications, and home-based exercise sessions on study. Participants receive supportive materials consisting of a Fitbit Aria scale, a Fitbit Charge 6 (or latest device), the Fitbit application (app), and access to the Cook for Your Life website on study. Participants also undergo blood sample collection on study.
  This arm includes participants who were randomized to ¡Vida! in Stage 1 and were responders (≥2% weight loss at 8 weeks).
  In Stage 2, responders receive additional ¡Vida! intervention programming.
  Interventions: Behavioral: ¡Vida! program
- Arm B - Stage 1: ¡Vida!; Stage 2: ¡Vida! + ¡Vida! Plus (Experimental): Participants participate in the online ¡Vida! program consisting of 24 health education online sessions, dietary modifications, and home-based exercise sessions on study. Participants receive supportive materials consisting of a Fitbit Aria scale, a Fitbit Charge 6 (or latest device), the Fitbit application (app), and access to the Cook for Your Life website on study. Participants also receive Experiential Learning (EL) by attending 14 remote lifestyle health education sessions. Participants also undergo blood sample collection on study.
  This arm includes participants who were randomized to ¡Vida! in Stage 1 and were non-responders (<2% weight loss at 8 weeks).
  In Stage 2, non-responders receive ¡Vida! Plus programming: the ¡Vida! Program plus Experiential Learning (EL).
  Interventions: Behavioral: ¡Vida! program; Behavioral: ¡Vida! Plus [¡Vida! + Experiential Learning (EL)]
- Arm C - Stage 1: ¡Vida!; Stage 2: ¡Vida! + ¡Vida! Plus + Health Coaching (HC) (Experimental): Participants participate in the online ¡Vida! program consisting of 24 health education online sessions, dietary modifications, and home-based exercise sessions on study. Participants receive supportive materials consisting of a Fitbit Aria scale, a Fitbit Charge 6 (or latest device), the Fitbit application (app), and access to the Cook for Your Life website on study. Participants also receive Experiential Learning (EL) by attending 14 remote lifestyle health education sessions. Participants also receive 9 30-minute individualized telephone health coaching sessions. Participants also undergo blood sample collection on study.
  This arm includes participants who were randomized to ¡Vida! in Stage 1 and were non-responders (<2% weight loss at 8 weeks).
  In Stage 2, non-responders receive ¡Vida! Plus programming: the ¡Vida! Program plus Experiential Learning (EL), and also receive health coaching.
  Interventions: Behavioral: ¡Vida! program; Behavioral: ¡Vida! Plus [¡Vida! + Experiential Learning (EL)]; Behavioral: Health Coaching
- Arm D - Stage 1: ¡Vida! + ¡Vida! Plus; Stage 2: ¡Vida! + ¡Vida! Plus (Experimental): Participants participate in the online ¡Vida! program consisting of 24 health education online sessions, dietary modifications, and home-based exercise sessions on study. Participants receive supportive materials consisting of a Fitbit Aria scale, a Fitbit Charge 6 (or latest device), the Fitbit application (app), and access to the Cook for Your Life website on study. Participants also receive Experiential Learning (EL) by attending 14 remote lifestyle health education sessions. Participants also undergo blood sample collection on study.
  This arm includes participants who were randomized to ¡Vida! + ¡Vida! Plus in Stage 1 and were responders (≥2% weight loss at 8 weeks).
  In Stage 2, responders receive additional ¡Vida! Plus intervention programming.
  Interventions: Behavioral: ¡Vida! program; Behavioral: ¡Vida! Plus [¡Vida! + Experiential Learning (EL)]
- Arm E - Stage 1: ¡Vida! + ¡Vida! Plus; Stage 2: ¡Vida! + ¡Vida! Plus + Health Coaching (HC) (Experimental): Participants participate in the online ¡Vida! program consisting of 24 health education online sessions, dietary modifications, and home-based exercise sessions on study. Participants receive supportive materials consisting of a Fitbit Aria scale, a Fitbit Charge 6 (or latest device), the Fitbit application (app), and access to the Cook for Your Life website on study. Participants also receive Experiential Learning (EL) by attending 14 remote lifestyle health education sessions. Participants also receive 9 30-minute individualized telephone health coaching sessions. Participants also undergo blood sample collection on study.
  This arm includes participants who were randomized to ¡Vida! + ¡Vida! Plus in Stage 1 and were non-responders (<2% weight loss at 8 weeks).
  In Stage 2, non-responders receive additional ¡Vida! Plus intervention programming, and also receive health coaching.
  Interventions: Behavioral: ¡Vida! program; Behavioral: ¡Vida! Plus [¡Vida! + Experiential Learning (EL)]; Behavioral: Health Coaching
- Arm F-Stage 1:¡Vida! + ¡Vida! Plus; Stage 2:¡Vida! + ¡Vida! Plus + Health Coaching + Mailed Toolkits (Experimental): Participants participate in the online ¡Vida! program consisting of 24 health education online sessions, dietary modifications, and home-based exercise sessions on study. Participants receive supportive materials consisting of a Fitbit Aria scale, a Fitbit Charge 6 (or latest device), the Fitbit application (app), and access to the Cook for Your Life website on study. Participants also receive Experiential Learning (EL) by attending 14 remote lifestyle health education sessions. Participants also receive 9 30-minute individualized telephone health coaching sessions, and receive a mailed toolkit of health items twice on study. Participants also undergo blood sample collection on study.
  This arm includes participants who were randomized to ¡Vida! + ¡Vida! Plus in Stage 1 and were non-responders (<2% weight loss at 8 weeks).
  In Stage 2, non-responders receive additional ¡Vida! Plus intervention programming, and also receive health coaching (HC) as well as mailed toolkits (MT).
  Interventions: Behavioral: ¡Vida! program; Behavioral: ¡Vida! Plus [¡Vida! + Experiential Learning (EL)]; Behavioral: Health Coaching; Behavioral: Mailed Toolkits

INTERVENTIONS:
Behavioral: ¡Vida! program — Participate in ¡Vida! program
  Other Names: Behavioral Intervention
Behavioral: ¡Vida! Plus [¡Vida! + Experiential Learning (EL)] — Participate in ¡Vida! Plus program
  Arms: Arm B - Stage 1: ¡Vida!; Stage 2: ¡Vida! + ¡Vida! Plus; Arm C - Stage 1: ¡Vida!; Stage 2: ¡Vida! + ¡Vida! Plus + Health Coaching (HC); Arm D - Stage 1: ¡Vida! + ¡Vida! Plus; Stage 2: ¡Vida! + ¡Vida! Plus; Arm E - Stage 1: ¡Vida! + ¡Vida! Plus; Stage 2: ¡Vida! + ¡Vida! Plus + Health Coaching (HC); Arm F-Stage 1:¡Vida! + ¡Vida! Plus; Stage 2:¡Vida! + ¡Vida! Plus + Health Coaching + Mailed Toolkits
Behavioral: Health Coaching — Receive health coaching
  Arms: Arm C - Stage 1: ¡Vida!; Stage 2: ¡Vida! + ¡Vida! Plus + Health Coaching (HC); Arm E - Stage 1: ¡Vida! + ¡Vida! Plus; Stage 2: ¡Vida! + ¡Vida! Plus + Health Coaching (HC); Arm F-Stage 1:¡Vida! + ¡Vida! Plus; Stage 2:¡Vida! + ¡Vida! Plus + Health Coaching + Mailed Toolkits
Behavioral: Mailed Toolkits — Receive a mailed toolkit of health items
  Arms: Arm F-Stage 1:¡Vida! + ¡Vida! Plus; Stage 2:¡Vida! + ¡Vida! Plus + Health Coaching + Mailed Toolkits

SUMMARY:
This clinical trial evaluates remotely delivered, community-aligned weight loss interventions in Latina breast cancer survivors. Breast cancer is the second leading cause of cancer death among women in the US. There are population differences in breast cancer mortality, based on specific risk factors, including obesity. Cancer is the leading cause of death among Latinos, and among Latinas, breast cancer is the leading cause of cancer death. An estimated 80% of Latinas in the United States have overweight/obesity, which is associated with poorer breast cancer outcomes. However, few, if any, effective interventions exist to promote and maintain weight loss in Latina breast cancer survivors. The development of an adaptive program that provides survivors with the support they need, as opposed to what is typically available, to improve breast cancer survivorship.

DETAILED DESCRIPTION:
OUTLINE: This sequential multiple assignment randomized trial (SMART) will test four different community-aligned 12-month adaptive weight loss interventions.

BASELINE: Participants receive written instructions and website link to complete surveys along with supportive materials including a measuring tape, Aria Bluetooth-enabled scale, and may receive an Actigraph accelerometer to be worn for 7 days at baseline. Participants also undergo blood sample collection at baseline.

STAGE ONE: Eligible participants from the baseline run-in are randomized to participate in Stage One. In Stage One, participants are randomized to one of two groups: ¡Vida! or ¡Vida! Plus.

STAGE TWO: Percent weight loss is measured at week 8. Women who lose ≥2% of their body weight at week 8 will be considered "Responders" and will continue with their original randomization assignment in Stage Two.

Women in the Stage One ¡Vida! group who lose <2% of their body weight will be re-randomized in Stage Two to receive either ¡Vida! Plus or ¡Vida! Plus + health coaching (HC). Women in the Stage One ¡Vida! Plus group who lose <2% of their body weight will be re-randomized in Stage Two to receive either ¡Vida! Plus + HC or ¡Vida! Plus + HC + mailed toolkits (MT).

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* Age >= 18 years
* Self-identifies Hispanic/Latina
* Able to read and write in Spanish and/or English
* Previous diagnosis of stage I-III BC within the past 5 years
* No evidence of current, recurrent, or metastatic disease
* 60 days post treatment, including chemotherapy, radiation therapy, and cancer-related surgery (NOTE: current allowed therapies include endocrine therapy, CDK4/6 inhibitors (e.g. palbociclib,ribociclib, abemaciclib), HER2-directed therapies (e.g., trastuzumab, neratinib), and monoclonal antibodies (e.g., pertuzumab, pembrolizumab); surgery for breast reconstruction is allowed during the trial)
* Body mass index (BMI) >= 27 kg/m^2 initially assessed via self-reported height and weight and confirmed prior to randomization via a tape measure and Bluetooth-enabled scale
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Willingness to participate in all study activities
* Access to phone for study contacts
* Access to internet to participate in the online program and to be able to sync study devices
* Successful completion of at-home baseline assessments prior to randomization

Exclusion Criteria:

* Body mass index (BMI) < 27 kg/m^2 at time of baseline data collection
* Diabetic with current use of insulin or sulfonylurea medications (note: current use of metformin is allowed)
* Use of glucagon-like peptide-1 (GLP1) receptor agonist medications reported at baseline
* Current use of cytotoxic chemotherapy medications (e.g., capecitabine) or drug-antibody conjugates (e.g., trastuzumab emtansine [T-DM1], trastuzumab deruxtecan [T-DXd])
* Major comorbidities or physical limitations that would preclude from healthy weight loss, reducing energy intake or engaging in PA
* Pregnant, breastfeeding, or planning to become pregnant during the study period
* Use of exogenous hormones for gender affirmation
* For stool sample collection only: Self-reported use of oral or intravenous antibiotics, antifungals, or anti-parasitics during the past 6 months
* For stool sample collection only: Presence of self-reported ileostomy or colostomy
* For stool sample collection only: Presence of self-reported inflammatory bowel diseases (e.g., Crohn's disease, ulcerative colitis)
* Anticipated major surgical procedure (e.g., hysterectomy) within 3 months after study registration. Breast reconstruction is allowed during study participation.
* Concurrent enrollment in another weight loss or physical activity trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) percent change | Baseline to 12 months
  Will be assessed by the percent of weight loss at month 12 and compared across the four embedded adaptive intervention (EAI) groups using the doubly robust estimator model.

SECONDARY OUTCOMES:
Body weight (kg) percent change as moderated by baseline characteristics | Baseline to 12 months
  Will be determined by whether EAI effectiveness is moderated by baseline patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No